CLINICAL TRIAL: NCT02562040
Title: Impact of Treatment of Mild Sleep-Disordered Breathing on Children's Health
Brief Title: Pediatric Adenotonsillectomy Trial for Snoring
Acronym: PATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University Hospitals Cleveland Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Michigan (Other); University of Texas Southwestern Medical Center (Other); University of Rochester (Other); Children's Hospital of The King's Daughters (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Redline, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P001798; 1U011HL125307-O1A1 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Sleep-Disordered Breathing
Keywords: Pediatrics; Primary Snoring; Adenotonsillectomy
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Watchful Waiting; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watchful Waiting with Supportive Care (Active Comparator): All Watchful Waiting with Supportive Care (WWSC) participants will receive information about healthy sleep habits for children and appropriate clinical referrals for management of co-morbidities.
  Interventions: Behavioral: Watchful Waiting with Supportive Care (WWSC)
- Early Adenotonsillectomy (Experimental): All Early Adenotonsillectomy (eAT) participants will receive information about healthy sleep habits for children, undergo adenotonsillectomy within 4 weeks of randomization and receive appropriate clinical referrals for management of co-morbidities
  Interventions: Procedure: Early Adenotonsillectomy (eAT)

INTERVENTIONS:
Procedure: Early Adenotonsillectomy (eAT) — Standard clinical adenotonsillectomy within 4 weeks post randomization in addition to information about healthy sleep habits for children and appropriate clinical referrals for management of co-morbidities.
  Arms: Early Adenotonsillectomy
Behavioral: Watchful Waiting with Supportive Care (WWSC) — Information about healthy sleep habits for children and appropriate clinical referrals for management of co-morbidities.
  Arms: Watchful Waiting with Supportive Care

SUMMARY:
The purpose of this study is to evaluate the effects of early adenotonsillectomy (eAT) on the behavior, sleep-disordered breathing symptoms and quality of life for children who snore, but do not have obstructive sleep apnea, as well as identify factors that moderate responses to the surgery. Half of participants will receive eAT, while the other half will be observed with watchful waiting and supportive care.

DETAILED DESCRIPTION:
Adenotonsillectomies are performed more than 500,000 times per year in the United States, and is the most common surgery performed under general anesthesia in children. The majority of surgeries are performed for obstructed breathing rather than for infection or other indications.

The role of adenotonsillectomy (AT) in improving the 7-month neurocognitive, behavioral and health outcomes of children with frank obstructive sleep apnea (OSA) was recently addressed in the Childhood Adenotonsillectomy Trial (CHAT). The results of this rigorous, multicenter, randomized controlled trial provided critically important data indicating that adenotonsillectomy compared to watchful waiting resulted in improved behavior, quality of life, sleep-disordered breathing (SDB) symptoms and polysomnographic parameters.

However, the Childhood Adenotonsillectomy Trial addressed the role of surgery in the minority of operative candidates who have frank obstructive sleep apnea, only one form of sleep disordered breathing on a spectrum that includes a more common phenotype, primary snoring (also termed mild sleep disordered breathing (MSDB)). Mild sleep disordered breathing is characterized by snoring without frank obstruction or gas exchange abnormalities, and has a population prevalence of about 10% in children. Since most surgeries for obstructed breathing are performed for mild sleep disordered breathing rather than obstructive sleep apnea, the next logical question is whether surgery is also effective in improving symptoms and health outcomes in this large group of children.

The Pediatric Adenotonsillectomy Trial for Snoring (PATS) intends to take advantage of a successful collaboration of leaders in sleep medicine, otolaryngology and clinical trials to efficiently leverage experiences from the CHAT trial to evaluate the role of adenotonsillectomy in children with mild sleep disordered breathing while also aiming to resolve uncertainties regarding management approaches for pediatric mild sleep disordered breathing by addressing several critical issues:

1. Assess outcomes important to children and their families, particularly patient-reported outcomes such as behavior, quality of life, and sleep disturbances.
2. Examine differences in treatment responses among children who are at increased risk for mild sleep disordered breathing, such as pre-school children, minorities, and children with asthma or obesity.
3. Evaluate health care utilization of children with mild sleep disordered breathing.
4. Assess moderating influences such as second hand smoke, insufficient sleep, socioeconomic status and family functioning
5. Examine longer term (12 month) outcomes that were not feasible in the Childhood Adenotonsillectomy Trial (CHAT).

These aims have substantial public health significance given the high morbidity of sleep disordered breathing in children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild sleep-disordered breathing (MSDB) defined as meeting all of the following criteria:

  * Caregiver report of habitual snoring that occurs most of the night on at least three nights per week, and has been present for at least three months (on average occurring > 3 nights per week or more half of sleep time) and
  * Centrally-scored polysomnogram (PSG) confirming an obstructive apnea index (OAI) <1/hour and apnea-hypopnea index (AHI) ≤3/hour and no oxygen saturation (SpO2) desaturation < 90% in conjunction with obstructive events, confirmed on PSG.
* Tonsillar hypertrophy ≥2 based on a standardized scale of 0-4.
* Deemed to be a candidate for AT by otolaryngologist (ENT) evaluation (i.e., no technical issues that would be a contraindication for surgery such as submucous cleft palate.)
* Primary indication for AT is nocturnal obstructive symptoms (i.e., not recurrent infections or other indications).

Exclusion Criteria:

* Previous tonsillectomy, including partial tonsillectomy
* Recurrent tonsillitis that merits prompt adenotonsillectomy (AT) per the American Academy of Otolaryngology-Head and Neck Surgery Clinical Practice Guidelines (i.e., ≥7 episodes/yr in the past year; ≥5 episodes/year over the past 2 years or ≥3 episodes/yr over the past 3 years.)
* Severe obesity (body mass index (BMI) z-score ≥3).
* Failure to thrive, defined as either height or weight being below the 5th percentile for age and gender.
* Severe chronic health conditions that might hamper participation or confound key variables under study, including but not limited to:

  * Severe cardiopulmonary disorders such as cystic fibrosis, and congenital heart disease.
  * Bleeding disorders
  * Sickle Cell Disease
  * Epilepsy requiring medication
  * Significant cardiac arrhythmia noted on PSG including: non-sustained ventricular tachycardia, atrial fibrillation, second degree atrioventricular block, sustained bradycardia, or sustained tachycardia.
  * Other severe chronic health problems such as diabetes, narcolepsy, and poorly controlled asthma.
  * Known genetic, craniofacial, neurological or psychiatric conditions likely to affect the airway, cognition or behavior;
  * Current use of psychotropic medication (other than medications for attention deficit hyperactivity disorder, hypnotics, antihypertensives, hypoglycemic agents including insulin, anticonvulsants, anticoagulants, or growth hormone.
  * Diagnosis of autism spectrum disorder.
  * Intellectual deficit or assigned to a self-contained classroom for all academic subjects.
  * History of severe developmental disability or Adaptive Behavior Assessment System (ABAS-3) score ≤60.
* Children/caregivers planning to move out of the area within the year.
* Children in foster care.
* Children/caregivers who do not speak English or Spanish well enough to complete the neurobehavioral measures.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 459 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Redline, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Rui Wang, PhD, Principal Investigator — Brigham and Women's Hospital; Susan L. Furth, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (7):
- United States (7):
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals-Case Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia

REFERENCES:
- [Background] Bhattacharyya N, Lin HW. Changes and consistencies in the epidemiology of pediatric adenotonsillar surgery, 1996-2006. Otolaryngol Head Neck Surg. 2010 Nov;143(5):680-4. doi: 10.1016/j.otohns.2010.06.918. PMID 20974339
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257
- [Background] Marcus CL, Moore RH, Rosen CL, Giordani B, Garetz SL, Taylor HG, Mitchell RB, Amin R, Katz ES, Arens R, Paruthi S, Muzumdar H, Gozal D, Thomas NH, Ware J, Beebe D, Snyder K, Elden L, Sprecher RC, Willging P, Jones D, Bent JP, Hoban T, Chervin RD, Ellenberg SS, Redline S; Childhood Adenotonsillectomy Trial (CHAT). A randomized trial of adenotonsillectomy for childhood sleep apnea. N Engl J Med. 2013 Jun 20;368(25):2366-76. doi: 10.1056/NEJMoa1215881. Epub 2013 May 21. PMID 23692173
- [Background] Standards and indications for cardiopulmonary sleep studies in children. American Thoracic Society. Am J Respir Crit Care Med. 1996 Feb;153(2):866-78. doi: 10.1164/ajrccm.153.2.8564147. No abstract available.
- [Background] Goodwin JL, Babar SI, Kaemingk KL, Rosen GM, Morgan WJ, Sherrill DL, Quan SF; Tucson Children's Assessment of Sleep Apnea Study. Symptoms related to sleep-disordered breathing in white and Hispanic children: the Tucson Children's Assessment of Sleep Apnea Study. Chest. 2003 Jul;124(1):196-203. doi: 10.1378/chest.124.1.196. PMID 12853523
- [Background] Mitchell RB, Pereira KD, Friedman NR. Sleep-disordered breathing in children: survey of current practice. Laryngoscope. 2006 Jun;116(6):956-8. doi: 10.1097/01.MLG.0000216413.22408.FD. PMID 16735907
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Ward SD, Sheldon SH, Shiffman RN, Lehmann C, Spruyt K; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):e714-55. doi: 10.1542/peds.2012-1672. Epub 2012 Aug 27. PMID 22926176
- [Background] Redline S, Tishler PV, Schluchter M, Aylor J, Clark K, Graham G. Risk factors for sleep-disordered breathing in children. Associations with obesity, race, and respiratory problems. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1527-32. doi: 10.1164/ajrccm.159.5.9809079. PMID 10228121
- [Background] Reuveni H, Simon T, Tal A, Elhayany A, Tarasiuk A. Health care services utilization in children with obstructive sleep apnea syndrome. Pediatrics. 2002 Jul;110(1 Pt 1):68-72. doi: 10.1542/peds.110.1.68. PMID 12093948
- [Background] Tarasiuk A, Simon T, Tal A, Reuveni H. Adenotonsillectomy in children with obstructive sleep apnea syndrome reduces health care utilization. Pediatrics. 2004 Feb;113(2):351-6. doi: 10.1542/peds.113.2.351. PMID 14754948
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Aurora RN, Zak RS, Karippot A, Lamm CI, Morgenthaler TI, Auerbach SH, Bista SR, Casey KR, Chowdhuri S, Kristo DA, Ramar K; American Academy of Sleep Medicine. Practice parameters for the respiratory indications for polysomnography in children. Sleep. 2011 Mar 1;34(3):379-88. doi: 10.1093/sleep/34.3.379. PMID 21359087
- [Background] Roland PS, Rosenfeld RM, Brooks LJ, Friedman NR, Jones J, Kim TW, Kuhar S, Mitchell RB, Seidman MD, Sheldon SH, Jones S, Robertson P; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: Polysomnography for sleep-disordered breathing prior to tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jul;145(1 Suppl):S1-15. doi: 10.1177/0194599811409837. Epub 2011 Jun 15. PMID 21676944
- [Background] Archbold KH, Pituch KJ, Panahi P, Chervin RD. Symptoms of sleep disturbances among children at two general pediatric clinics. J Pediatr. 2002 Jan;140(1):97-102. doi: 10.1067/mpd.2002.119990. PMID 11815771
- [Background] O'Brien LM, Holbrook CR, Mervis CB, Klaus CJ, Bruner JL, Raffield TJ, Rutherford J, Mehl RC, Wang M, Tuell A, Hume BC, Gozal D. Sleep and neurobehavioral characteristics of 5- to 7-year-old children with parentally reported symptoms of attention-deficit/hyperactivity disorder. Pediatrics. 2003 Mar;111(3):554-63. doi: 10.1542/peds.111.3.554. PMID 12612236
- [Background] Greenfeld M, Sivan Y, Tauman R. The effect of seasonality on sleep-disordered breathing severity in children. Sleep Med. 2013 Oct;14(10):991-4. doi: 10.1016/j.sleep.2013.03.026. Epub 2013 Jul 25. PMID 23890953
- [Background] Boss EF, Marsteller JA, Simon AE. Outpatient tonsillectomy in children: demographic and geographic variation in the United States, 2006. J Pediatr. 2012 May;160(5):814-9. doi: 10.1016/j.jpeds.2011.11.041. Epub 2011 Dec 17. PMID 22183449
- [Background] Friedman NR, Perkins JN, McNair B, Mitchell RB. Current practice patterns for sleep-disordered breathing in children. Laryngoscope. 2013 Apr;123(4):1055-8. doi: 10.1002/lary.23709. Epub 2013 Feb 4. PMID 23382017
- [Background] Morrell MJ, Finn L, Kim H, Peppard PE, Badr MS, Young T. Sleep fragmentation, awake blood pressure, and sleep-disordered breathing in a population-based study. Am J Respir Crit Care Med. 2000 Dec;162(6):2091-6. doi: 10.1164/ajrccm.162.6.9904008. PMID 11112120
- [Background] Teodorescu M, Polomis DA, Hall SV, Teodorescu MC, Gangnon RE, Peterson AG, Xie A, Sorkness CA, Jarjour NN. Association of obstructive sleep apnea risk with asthma control in adults. Chest. 2010 Sep;138(3):543-50. doi: 10.1378/chest.09-3066. Epub 2010 May 21. PMID 20495105
- [Background] Teodorescu M, Polomis DA, Teodorescu MC, Gangnon RE, Peterson AG, Consens FB, Chervin RD, Jarjour NN. Association of obstructive sleep apnea risk or diagnosis with daytime asthma in adults. J Asthma. 2012 Aug;49(6):620-8. doi: 10.3109/02770903.2012.689408. Epub 2012 Jun 28. PMID 22742082
- [Background] Horne RS, Yang JS, Walter LM, Richardson HL, O'Driscoll DM, Foster AM, Wong S, Ng ML, Bashir F, Patterson R, Nixon GM, Jolley D, Walker AM, Anderson V, Trinder J, Davey MJ. Elevated blood pressure during sleep and wake in children with sleep-disordered breathing. Pediatrics. 2011 Jul;128(1):e85-92. doi: 10.1542/peds.2010-3431. Epub 2011 Jun 27. PMID 21708802
- [Background] Chervin RD, Ruzicka DL, Giordani BJ, Weatherly RA, Dillon JE, Hodges EK, Marcus CL, Guire KE. Sleep-disordered breathing, behavior, and cognition in children before and after adenotonsillectomy. Pediatrics. 2006 Apr;117(4):e769-78. doi: 10.1542/peds.2005-1837. PMID 16585288
- [Background] Ross KR, Storfer-Isser A, Hart MA, Kibler AM, Rueschman M, Rosen CL, Kercsmar CM, Redline S. Sleep-disordered breathing is associated with asthma severity in children. J Pediatr. 2012 May;160(5):736-42. doi: 10.1016/j.jpeds.2011.10.008. Epub 2011 Dec 1. PMID 22133422
- [Background] Friberg D, Ansved T, Borg K, Carlsson-Nordlander B, Larsson H, Svanborg E. Histological indications of a progressive snorers disease in an upper airway muscle. Am J Respir Crit Care Med. 1998 Feb;157(2):586-93. doi: 10.1164/ajrccm.157.2.96-06049. PMID 9476877
- [Background] Friberg D, Gazelius B, Hokfelt T, Nordlander B. Abnormal afferent nerve endings in the soft palatal mucosa of sleep apnoics and habitual snorers. Regul Pept. 1997 Jul 23;71(1):29-36. doi: 10.1016/s0167-0115(97)01016-1. PMID 9299639
- [Background] Bergeron C, Kimoff J, Hamid Q. Obstructive sleep apnea syndrome and inflammation. J Allergy Clin Immunol. 2005 Dec;116(6):1393-6. doi: 10.1016/j.jaci.2005.10.008. No abstract available. PMID 16337480
- [Background] Devouassoux G, Levy P, Rossini E, Pin I, Fior-Gozlan M, Henry M, Seigneurin D, Pepin JL. Sleep apnea is associated with bronchial inflammation and continuous positive airway pressure-induced airway hyperresponsiveness. J Allergy Clin Immunol. 2007 Mar;119(3):597-603. doi: 10.1016/j.jaci.2006.11.638. Epub 2007 Jan 29. PMID 17261329
- [Background] Salerno FG, Carpagnano E, Guido P, Bonsignore MR, Roberti A, Aliani M, Vignola AM, Spanevello A. Airway inflammation in patients affected by obstructive sleep apnea syndrome. Respir Med. 2004 Jan;98(1):25-8. doi: 10.1016/j.rmed.2003.08.003. PMID 14959810
- [Background] Lee SA, Amis TC, Byth K, Larcos G, Kairaitis K, Robinson TD, Wheatley JR. Heavy snoring as a cause of carotid artery atherosclerosis. Sleep. 2008 Sep;31(9):1207-13. PMID 18788645
- [Background] Kingshott RN, Engleman HM, Deary IJ, Douglas NJ. Does arousal frequency predict daytime function? Eur Respir J. 1998 Dec;12(6):1264-70. doi: 10.1183/09031936.98.12061264. PMID 9877475
- [Background] Blunden S, Lushington K, Kennedy D, Martin J, Dawson D. Behavior and neurocognitive performance in children aged 5-10 years who snore compared to controls. J Clin Exp Neuropsychol. 2000 Oct;22(5):554-68. doi: 10.1076/1380-3395(200010)22:5;1-9;FT554. PMID 11094391
- [Background] O'Brien LM, Mervis CB, Holbrook CR, Bruner JL, Klaus CJ, Rutherford J, Raffield TJ, Gozal D. Neurobehavioral implications of habitual snoring in children. Pediatrics. 2004 Jul;114(1):44-9. doi: 10.1542/peds.114.1.44. PMID 15231906
- [Background] Melendres MC, Lutz JM, Rubin ED, Marcus CL. Daytime sleepiness and hyperactivity in children with suspected sleep-disordered breathing. Pediatrics. 2004 Sep;114(3):768-75. doi: 10.1542/peds.2004-0730. PMID 15342852
- [Background] Emancipator JL, Storfer-Isser A, Taylor HG, Rosen CL, Kirchner HL, Johnson NL, Zambito AM, Redline S. Variation of cognition and achievement with sleep-disordered breathing in full-term and preterm children. Arch Pediatr Adolesc Med. 2006 Feb;160(2):203-10. doi: 10.1001/archpedi.160.2.203. PMID 16461879
- [Background] Robertson A, Johnson P, Middleton S, Norman M, Hennessy A. PP155. Relationship between overnight blood pressure and snoring during pregnancy. Pregnancy Hypertens. 2012 Jul;2(3):322-3. doi: 10.1016/j.preghy.2012.04.266. Epub 2012 Jun 13. PMID 26105476
- [Background] Blyton DM, Skilton MR, Edwards N, Hennessy A, Celermajer DS, Sullivan CE. Treatment of sleep disordered breathing reverses low fetal activity levels in preeclampsia. Sleep. 2013 Jan 1;36(1):15-21. doi: 10.5665/sleep.2292. PMID 23288967
- [Background] Leupe P, Hox V, Debruyne F, Schrooten W, Claes NV, Lemkens N, Lemkens P. Tonsillectomy compared to acute tonsillitis in children: a comparison study of societal costs. B-ENT. 2012;8(2):103-11. PMID 22896929
- [Background] Pratt LW, Gallagher RA. Tonsillectomy and adenoidectomy: incidence and mortality, 1968--1972. Otolaryngol Head Neck Surg (1979). 1979 Mar-Apr;87(2):159-66. doi: 10.1177/019459987908700201. PMID 503482
- [Background] Tarasiuk A, Greenberg-Dotan S, Brin YS, Simon T, Tal A, Reuveni H. Determinants affecting health-care utilization in obstructive sleep apnea syndrome patients. Chest. 2005 Sep;128(3):1310-4. doi: 10.1378/chest.128.3.1310. PMID 16162723
- [Background] Rasch B, Born J. About sleep's role in memory. Physiol Rev. 2013 Apr;93(2):681-766. doi: 10.1152/physrev.00032.2012. PMID 23589831
- [Background] Redline S, Tishler PV, Hans MG, Tosteson TD, Strohl KP, Spry K. Racial differences in sleep-disordered breathing in African-Americans and Caucasians. Am J Respir Crit Care Med. 1997 Jan;155(1):186-92. doi: 10.1164/ajrccm.155.1.9001310.
- [Background] Rosen CL, Larkin EK, Kirchner HL, Emancipator JL, Bivins SF, Surovec SA, Martin RJ, Redline S. Prevalence and risk factors for sleep-disordered breathing in 8- to 11-year-old children: association with race and prematurity. J Pediatr. 2003 Apr;142(4):383-9. doi: 10.1067/mpd.2003.28. PMID 12712055
- [Background] Ancoli-Israel S, Klauber MR, Stepnowsky C, Estline E, Chinn A, Fell R. Sleep-disordered breathing in African-American elderly. Am J Respir Crit Care Med. 1995 Dec;152(6 Pt 1):1946-9. doi: 10.1164/ajrccm.152.6.8520760.
- [Background] Montgomery-Downs HE, Jones VF, Molfese VJ, Gozal D. Snoring in preschoolers: associations with sleepiness, ethnicity, and learning. Clin Pediatr (Phila). 2003 Oct;42(8):719-26. doi: 10.1177/000992280304200808. PMID 14601921
- [Background] Friedman M, Bliznikas D, Klein M, Duggal P, Somenek M, Joseph NJ. Comparison of the incidences of obstructive sleep apnea-hypopnea syndrome in African-Americans versus Caucasian-Americans. Otolaryngol Head Neck Surg. 2006 Apr;134(4):545-50. doi: 10.1016/j.otohns.2005.12.011. PMID 16564370
- [Background] Kum-Nji P, Mangrem CL, Wells PJ, Klesges LM, Herrod HG. Black/white differential use of health services by young children in a rural Mississippi community. South Med J. 2006 Sep;99(9):957-62. doi: 10.1097/01.smj.0000232966.81950.a4. PMID 17004530
- [Background] Morton S, Rosen C, Larkin E, Tishler P, Aylor J, Redline S. Predictors of sleep-disordered breathing in children with a history of tonsillectomy and/or adenoidectomy. Sleep. 2001 Nov 1;24(7):823-9. doi: 10.1093/sleep/24.7.823. PMID 11683485
- [Background] Thongyam A, Marcus CL, Lockman JL, Cornaglia MA, Caroff A, Gallagher PR, Shults J, Traylor JT, Rizzi MD, Elden L. Predictors of perioperative complications in higher risk children after adenotonsillectomy for obstructive sleep apnea: a prospective study. Otolaryngol Head Neck Surg. 2014 Dec;151(6):1046-54. doi: 10.1177/0194599814552059. Epub 2014 Oct 9. PMID 25301788
- [Background] McLaughlin Crabtree V, Beal Korhonen J, Montgomery-Downs HE, Faye Jones V, O'Brien LM, Gozal D. Cultural influences on the bedtime behaviors of young children. Sleep Med. 2005 Jul;6(4):319-24. doi: 10.1016/j.sleep.2005.02.001. Epub 2005 Apr 1. PMID 15978515
- [Background] Cornelius LJ. Health habits of school-age children. J Health Care Poor Underserved. 1991 Winter;2(3):374-95. doi: 10.1353/hpu.2010.0414. PMID 1772949
- [Background] Vriend JL, Davidson FD, Corkum PV, Rusak B, Chambers CT, McLaughlin EN. Manipulating sleep duration alters emotional functioning and cognitive performance in children. J Pediatr Psychol. 2013 Nov;38(10):1058-69. doi: 10.1093/jpepsy/jst033. Epub 2013 May 28. PMID 23720415
- [Background] Spilsbury JC, Storfer-Isser A, Kirchner HL, Nelson L, Rosen CL, Drotar D, Redline S. Neighborhood disadvantage as a risk factor for pediatric obstructive sleep apnea. J Pediatr. 2006 Sep;149(3):342-7. doi: 10.1016/j.jpeds.2006.04.061. PMID 16939744
- [Background] Sulit LG, Storfer-Isser A, Rosen CL, Kirchner HL, Redline S. Associations of obesity, sleep-disordered breathing, and wheezing in children. Am J Respir Crit Care Med. 2005 Mar 15;171(6):659-64. doi: 10.1164/rccm.200403-398OC. Epub 2004 Dec 10. PMID 15591475
- [Background] Ersu R, Arman AR, Save D, Karadag B, Karakoc F, Berkem M, Dagli E. Prevalence of snoring and symptoms of sleep-disordered breathing in primary school children in istanbul. Chest. 2004 Jul;126(1):19-24. doi: 10.1378/chest.126.1.19. PMID 15249437
- [Background] Kaditis AG, Kalampouka E, Hatzinikolaou S, Lianou L, Papaefthimiou M, Gartagani-Panagiotopoulou P, Zintzaras E, Chrousos G. Associations of tonsillar hypertrophy and snoring with history of wheezing in childhood. Pediatr Pulmonol. 2010 Mar;45(3):275-80. doi: 10.1002/ppul.21174. PMID 20131382
- [Background] Li AM, Au CT, So HK, Lau J, Ng PC, Wing YK. Prevalence and risk factors of habitual snoring in primary school children. Chest. 2010 Sep;138(3):519-27. doi: 10.1378/chest.09-1926. Epub 2010 Feb 19. PMID 20173057
- [Background] Marshall NS, Almqvist C, Grunstein RR, Marks GB; Childhood Asthma Prevention Study. Predictors for snoring in children with rhinitis at age 5. Pediatr Pulmonol. 2007 Jul;42(7):584-91. doi: 10.1002/ppul.20606. PMID 17534968
- [Background] Kuehni CE, Strippoli MP, Chauliac ES, Silverman M. Snoring in preschool children: prevalence, severity and risk factors. Eur Respir J. 2008 Feb;31(2):326-33. doi: 10.1183/09031936.00088407. Epub 2007 Nov 21. PMID 18032441
- [Background] Kheirandish-Gozal L, Dayyat EA, Eid NS, Morton RL, Gozal D. Obstructive sleep apnea in poorly controlled asthmatic children: effect of adenotonsillectomy. Pediatr Pulmonol. 2011 Sep;46(9):913-8. doi: 10.1002/ppul.21451. Epub 2011 Apr 4. PMID 21465680
- [Background] Bloom B, Cohen RA, Freeman G. Summary health statistics for U.S. children: National Health Interview Survey, 2010. Vital Health Stat 10. 2011 Dec;(250):1-80. PMID 22338334
- [Background] Kaditis AG, Finder J, Alexopoulos EI, Starantzis K, Tanou K, Gampeta S, Agorogiannis E, Christodoulou S, Pantazidou A, Gourgoulianis K, Molyvdas PA. Sleep-disordered breathing in 3,680 Greek children. Pediatr Pulmonol. 2004 Jun;37(6):499-509. doi: 10.1002/ppul.20002. PMID 15114550
- [Background] Corbo GM, Fuciarelli F, Foresi A, De Benedetto F. Snoring in children: association with respiratory symptoms and passive smoking. BMJ. 1989 Dec 16;299(6714):1491-4. doi: 10.1136/bmj.299.6714.1491. PMID 2514859
- [Background] Weinstock TG, Rosen CL, Marcus CL, Garetz S, Mitchell RB, Amin R, Paruthi S, Katz E, Arens R, Weng J, Ross K, Chervin RD, Ellenberg S, Wang R, Redline S. Predictors of obstructive sleep apnea severity in adenotonsillectomy candidates. Sleep. 2014 Feb 1;37(2):261-9. doi: 10.5665/sleep.3394. PMID 24497655
- [Background] Richards W, Ferdman RM. Prolonged morbidity due to delays in the diagnosis and treatment of obstructive sleep apnea in children. Clin Pediatr (Phila). 2000 Feb;39(2):103-8. doi: 10.1177/000992280003900205. PMID 10696547
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Aickin M, Gensler H. Adjusting for multiple testing when reporting research results: the Bonferroni vs Holm methods. Am J Public Health. 1996 May;86(5):726-8. doi: 10.2105/ajph.86.5.726. PMID 8629727
- [Background] Gottlieb DJ, Chase C, Vezina RM, Heeren TC, Corwin MJ, Auerbach SH, Weese-Mayer DE, Lesko SM. Sleep-disordered breathing symptoms are associated with poorer cognitive function in 5-year-old children. J Pediatr. 2004 Oct;145(4):458-64. doi: 10.1016/j.jpeds.2004.05.039. PMID 15480367
- [Background] Orchinik LJ, Taylor HG, Espy KA, Minich N, Klein N, Sheffield T, Hack M. Cognitive outcomes for extremely preterm/extremely low birth weight children in kindergarten. J Int Neuropsychol Soc. 2011 Nov;17(6):1067-79. doi: 10.1017/S135561771100107X. Epub 2011 Sep 19. PMID 21923973
- [Background] Fritz MS, Mackinnon DP. Required sample size to detect the mediated effect. Psychol Sci. 2007 Mar;18(3):233-9. doi: 10.1111/j.1467-9280.2007.01882.x. PMID 17444920
- [Background] MacKinnon DP, Fritz MS, Williams J, Lockwood CM. Distribution of the product confidence limits for the indirect effect: program PRODCLIN. Behav Res Methods. 2007 Aug;39(3):384-9. doi: 10.3758/bf03193007. PMID 17958149
- [Background] White IR, Royston P, Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. Stat Med. 2011 Feb 20;30(4):377-99. doi: 10.1002/sim.4067. Epub 2010 Nov 30. PMID 21225900
- [Background] Bang H, Robins JM. Doubly robust estimation in missing data and causal inference models. Biometrics. 2005 Dec;61(4):962-73. doi: 10.1111/j.1541-0420.2005.00377.x. PMID 16401269
- [Background] Zhao L, Tian L, Cai T, Claggett B, Wei LJ. EFFECTIVELY SELECTING A TARGET POPULATION FOR A FUTURE COMPARATIVE STUDY. J Am Stat Assoc. 2013 Jan 1;108(502):527-539. doi: 10.1080/01621459.2013.770705. PMID 24058223
- [Background] Foster JC, Taylor JM, Ruberg SJ. Subgroup identification from randomized clinical trial data. Stat Med. 2011 Oct 30;30(24):2867-80. doi: 10.1002/sim.4322. Epub 2011 Aug 4. PMID 21815180
- [Background] Haybittle JL. Repeated assessment of results in clinical trials of cancer treatment. Br J Radiol. 1971 Oct;44(526):793-7. doi: 10.1259/0007-1285-44-526-793. No abstract available. PMID 4940475
- [Background] Peto R, Pike MC, Armitage P, Breslow NE, Cox DR, Howard SV, Mantel N, McPherson K, Peto J, Smith PG. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. I. Introduction and design. Br J Cancer. 1976 Dec;34(6):585-612. doi: 10.1038/bjc.1976.220. PMID 795448
- [Derived] Gong W, Huang K, Psychogios I, Li S, Chen L, Zhang J, Fang F, Zhang Z, Hu Y. Growth and sleep outcomes after adenotonsillectomy in pediatric mild sleep-disordered breathing. Sci Rep. 2025 Dec 5;16(1):688. doi: 10.1038/s41598-025-30271-3. PMID 41350327
- [Derived] Cabrera AJ, Li D, Redline S, Chervin RD, Ishman SL, Baldassari CM, Mitchell RB, Amin R, Hassan F, Ibrahim S, Ross KR, Kirkham EM, Zopf DA, Cielo CM, Young LR, Furth SL, Garetz S, Rosen CL, Wang R, Tapia IE. Adenotonsillectomy and Blood Pressure in Children With Mild Obstructive Sleep-Disordered Breathing: An Exploratory Analysis of the PATS Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Oct 1;151(10):957-966. doi: 10.1001/jamaoto.2025.2555. PMID 40875240
- [Derived] Bakker JP, Zhang F, Amin R, Baldassari CM, Chervin RD, Garetz SL, Hassan F, Ibrahim S, Ishman SL, Kirkham EM, Linden A, Mitchell RB, Naqvi K, Rosen CL, Ross K, Tapia IE, Young LR, Yu PK, Redline S, Wang R. Adenotonsillectomy and Health Care Utilization in Children With Snoring and Mild Sleep Apnea: A Randomized Clinical Trial. JAMA Pediatr. 2025 Jun 1;179(6):600-609. doi: 10.1001/jamapediatrics.2025.0023. PMID 40094698
- [Derived] Tsou PY, Gueye-Ndiaye S, Gorman KL, Williamson A, Ibrahim S, Weber S, Zopf D, Hassan F, Baldassari C, Sendon C, Wang R, Redline S, Li D, Ross KR. Asthma and sleep disordered breathing in the pediatric adenotonsillectomy trial for snoring study. Sleep Breath. 2024 Dec 4;29(1):46. doi: 10.1007/s11325-024-03210-1. PMID 39633037
- [Derived] Ibrahim S, Ievers-Landis CE, Taylor HG, Tapia IE, Williamson AA, Cole MC, Gurbani N, Chervin RD, Hassan F, Mitchell RB, Naqvi K, Baldassari C, Edlund W, Wang R, Wei Z, Li D, Redline S, Rosen CL. Bedsharing sleep characteristics in children with mild sleep-disordered breathing. J Clin Sleep Med. 2025 Feb 1;21(2):237-247. doi: 10.5664/jcsm.11352. PMID 39302128
- [Derived] Kirkham EM, Ishman S, Baldassari CM, Mitchell RB, Naqvi SK, Tapia IE, Elden LM, Hassan F, Ibrahim S, Ross K, Cen M, Wang R, Redline S, Chervin RD. Weight Gain After Adenotonsillectomy in Children With Mild Obstructive Sleep-Disordered Breathing: Exploratory Analysis of the PATS Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Oct 1;150(10):859-867. doi: 10.1001/jamaoto.2024.2554. PMID 39172463
- [Derived] Gueye-Ndiaye S, Tully M, Amin R, Baldassari CM, Chervin RD, Cole M, Ibrahim S, Kirkham EM, Mitchell RB, Naqvi K, Ross K, Rueschman M, Tapia IE, Williamson AA, Wei Z, Rosen CL, Wang R, Redline S. Neighborhood Disadvantage, Quality of Life, and Symptom Burden in Children with Mild Sleep-disordered Breathing. Ann Am Thorac Soc. 2024 Apr;21(4):604-611. doi: 10.1513/AnnalsATS.202307-653OC. PMID 38241286
- [Derived] Mitchell RB, Cook K, Garetz S, Tapia IE, Elden LM, Kirkham EM, Shah J, Otteson T, Zopf D, Amin R, Ishman S, Baldassari CM, Chervin RD, Hassan F, Naqvi K, Wang R, Redline S. Clinical Characteristics of Primary Snoring vs Mild Obstructive Sleep Apnea in Children: Analysis of the Pediatric Adenotonsillectomy for Snoring (PATS) Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Feb 1;150(2):99-106. doi: 10.1001/jamaoto.2023.3816. PMID 38095903
- [Derived] Redline S, Cook K, Chervin RD, Ishman S, Baldassari CM, Mitchell RB, Tapia IE, Amin R, Hassan F, Ibrahim S, Ross K, Elden LM, Kirkham EM, Zopf D, Shah J, Otteson T, Naqvi K, Owens J, Young L, Furth S, Connolly H, Clark CAC, Bakker JP, Garetz S, Radcliffe J, Taylor HG, Rosen CL, Wang R; Pediatric Adenotonsillectomy Trial for Snoring (PATS) Study Team. Adenotonsillectomy for Snoring and Mild Sleep Apnea in Children: A Randomized Clinical Trial. JAMA. 2023 Dec 5;330(21):2084-2095. doi: 10.1001/jama.2023.22114. PMID 38051326
- [Derived] Robinson KA, Wei Z, Radcliffe J, Taylor HG, Baldassari CM, Chervin RD, Ishman S, Mitchell RB, Tapia IE, Garetz S, Hassan F, Ibrahim S, Elden LM, Ievers-Landis CE, Williamson AA, Hjelm M, Kirkham E, Tham A, Naqvi K, Rueschman M, Rosen CL, Wang R, Redline S. Associations of actigraphy measures of sleep duration and continuity with executive function, vigilance, and fine motor control in children with snoring and mild sleep-disordered breathing. J Clin Sleep Med. 2023 Sep 1;19(9):1595-1603. doi: 10.5664/jcsm.10620. PMID 37185231
- [Derived] Clark CAC, Cook K, Wang R, Rueschman M, Radcliffe J, Redline S, Taylor HG. Psychometric properties of a combined go/no-go and continuous performance task across childhood. Psychol Assess. 2023 Apr;35(4):353-365. doi: 10.1037/pas0001202. Epub 2023 Jan 12. PMID 36633982
- [Derived] Yu PK, Radcliffe J, Gerry Taylor H, Amin RS, Baldassari CM, Boswick T, Chervin RD, Elden LM, Furth SL, Garetz SL, George A, Ishman SL, Kirkham EM, Liu C, Mitchell RB, Kamal Naqvi S, Rosen CL, Ross KR, Shah JR, Tapia IE, Young LR, Zopf DA, Wang R, Redline S. Neurobehavioral morbidity of pediatric mild sleep-disordered breathing and obstructive sleep apnea. Sleep. 2022 May 12;45(5):zsac035. doi: 10.1093/sleep/zsac035. Epub 2022 Feb 12. PMID 35554583
- [Derived] Wang R, Bakker JP, Chervin RD, Garetz SL, Hassan F, Ishman SL, Mitchell RB, Morrical MG, Naqvi SK, Radcliffe J, Riggan EI, Rosen CL, Ross K, Rueschman M, Tapia IE, Taylor HG, Zopf DA, Redline S. Pediatric Adenotonsillectomy Trial for Snoring (PATS): protocol for a randomised controlled trial to evaluate the effect of adenotonsillectomy in treating mild obstructive sleep-disordered breathing. BMJ Open. 2020 Mar 15;10(3):e033889. doi: 10.1136/bmjopen-2019-033889. PMID 32179560

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Started | 228 | 231
6-month Visit | 189 | 188
Completed | 199 (Of the 199 subjects that completed the final 12-month visit; 178 had baseline, 6-month and 12-month visits, and 21 had only baseline and 12-month visits) | 196 (Of the 196 subjects that completed the final 12-month visit; 177 had baseline, 6-month and 12-month visits, and 19 had only baseline and 12-month visits)
Not Completed | 29 | 35
Not completed — Lost to Follow-up | 20 | 28
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy | Total
Number analyzed (Participants) | 227 | 231 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Primary analysis includes all PATS participants other than one child who was randomized from Boston Children's Hospital (site's only participant was lost to follow-up and site closed early)
  years | 6.15 (2.36) | 6.10 (2.25) | 6.13 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Primary analysis includes all PATS participants other than one child who was randomized from Boston Children's Hospital (site's only participant was lost to follow-up and site closed early)
  Participants
    Female | 111 | 119 | 230
    Male | 116 | 112 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Primary analysis includes all PATS participants other than one child who was randomized from Boston Children's Hospital (site's only participant was lost to follow-up and site closed early)
  Participants
    Hispanic or Latino | 33 | 42 | 75
    Not Hispanic or Latino | 194 | 189 | 383
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Primary analysis includes all PATS participants other than one child who was randomized from Boston Children's Hospital (site's only participant was lost to follow-up and site closed early)
  Participants
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 5 | 3 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 63 | 60 | 123
    White | 148 | 155 | 303
    More than one race | 10 | 10 | 20
    Unknown or Not Reported | 0 | 1 | 1
Apnea-Hypopnea Index [Median (Inter-Quartile Range); unit: events per hour] — Sum of all obstructive apneas, mixed apneas, and hypopneas associated with oxygen desaturations >=3% and/or arousal; divided by total sleep time in hours, to create an hourly rate. Population: Primary analysis includes all PATS participants other than one child who was randomized from Boston Children's Hospital (site's only participant was lost to follow-up and site closed early)
  events per hour | 0.6 [0.3 to 1.15] | 0.5 [0.1 to 1.1] | 0.5 [0.2 to 1.1]
Asthma [Count of Participants; unit: Participants] — Diagnosed by a medical professional Population: Primary analysis includes all PATS participants other than one child who was randomized from Boston Children's Hospital (site's only participant was lost to follow-up and site closed early)
  Participants | 55 | 53 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Months in Caregiver-reported Behavior Rating Inventory of Executive Function (BRIEF) Global Executive Composite (GEC) T Score
Description: The BRIEF GEC section comprises summary measures of behavioral regulation, emotion regulation, and cognitive regulation (BRIEF-2, for children aged 5 to 18 years) or inhibitory self-control, flexibility, and emergent metacognition (BRIEF-P, for preschool-aged children). These scores are linear transformations of the raw scores (mean = 50, sd = 10) where a higher T score indicates a child has a lower capacity to organize and self-regulate.
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 197 | 195
change in score on a scale | -1.90 (8.62) | -3.08 (9.39)

2. Primary Outcome: Change From Baseline to 12 Months in Go-No-Go (GNG) Signal Detection Parameter D-prime (d').
Description: Performance on combined Go-No-Go (GNG)/Continuous Performance Test (CPT) task was assessed by tracking accuracy responses to targets (fish) and false positive responses to non-targets (sharks). d' is computed for both portions of the task as an assessment of accuracy in making correct detections adjusting for the participant's tendency to respond to non-targets. The adjusted measure is computed by subtracting Z-scores for false positive responses from Z-scores for correct detections. Individual Z-scores were based on a child's performance within same age groups (3-4, 5-6 , and >=7 years old). Scores ranged across age groups from -0.53 to 3.99 for GNG and -0.61 to 4.35 for CPT. Higher scores reflect better discrimination of targets from non-targets. A value of 4.65 represents 100% accuracy, 0 represents chance performance, and minus scores represent more frequent detection of non-targets than targets, suggesting a child misunderstood instructions or preferred responding to non-targets.
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: d-prime
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 182 | 182
d-prime | 1.9 (8.6) | 3.1 (9.4)

3. Secondary Outcome: Change From Baseline to 12 Months in NIH-Toolbox 9-Hole Pegboard Dexterity Test Time
Description: Fine motor coordination assessed by the time (in seconds) it takes a child to complete the NIH-Toolbox 9-Hole Pegboard Dexterity Test. Shorter times indicate greater dexterity. The reported value is the average of the dominant and non-dominant hand scores.
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in seconds
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 183 | 187
change in seconds | -5.9 (8.0) | -5.3 (7.4)

4. Secondary Outcome: Change From Baseline to 12 Months in Child Behavior Checklist (CBCL) Summary Scale T Scores
Description: Behavior assessed by the change from baseline to 12 months in the caregiver-reported Child Behavior Checklist (CBCL) overall summary score T scores. The T scores are standardized transformations of the raw score (mean = 50, sd = 10), where a higher scores indicate greater problems.
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 182 | 183
change in score on a scale | -1.44 (7.54) | -4.55 (9.00)

5. Secondary Outcome: Change From Baseline to 12 Months in Pediatric Sleep Questionnaire: Sleep-Related Breathing Disorder Scale (PSQ-SRBD) Total Score.
Description: The PSQ-SRBD scale is a 22-item questionnaire which includes three subscales: snoring, daytime sleepiness, and hyperactive behaviors/inattention. The PSQ-SRBD is commonly used to assess sleep-disordered breathing (SDB) risk in pediatric patients, but is also increasingly used to assess symptom burden. Higher scores correspond to greater SDB symptoms and the total range is 0-1
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 193 | 187
change in score on a scale | -0.07 (0.16) | -0.23 (0.19)

6. Secondary Outcome: Change From Baseline to 12 Months in Sleepiness Measured by Change in the Epworth Sleepiness Scale (ESS) Modified for Children Summary Score.
Description: The Epworth Sleepiness Scale (ESS) Modified for Children is an 8-item validated questionnaire which evaluates excessive daytime sleepiness. The wording and questions are revised from the original ESS to be more suitable for children. The total score has a range from 0-24 where higher values indicate greater sleepiness.
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 193 | 184
change in score on a scale | -0.67 (4.39) | -1.77 (4.95)

7. Secondary Outcome: Change From Baseline to 12 Months in Pediatric Quality of Life Inventory (PedsQL) Caregiver Reported Total Score and Subscales.
Description: General quality of life assessed by caregiver reported PedsQL total score and subscores (Psychosocial Health Summary Score & Physical Health Summary Score). The PedsQL Total Score comprises performance on 4 subscales: emotional functioning, social functioning, school functioning (summarized by the Psychosocial Functioning Score) and physical functioning (summarized by the Physical Functioning score). Scores on all scales range from 0 to 100, with higher scores indicating an increased quality of life.
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 193 | 187
change in score on a scale
  Parent - Total | -2.62 (15.02) | 2.09 (14.95)
  Parent - Physical | -5.34 (24.32) | 0.74 (23.55)
  Parent - Psychosocial | -1.08 (13.33) | 2.85 (14.17)

8. Secondary Outcome: Change From Baseline to 12 Months in Quality of Life Survey Evaluation of Sleep-Disordered Breathing (OSA-18) Total Score.
Description: The OSA-18 is a disease-specific QOL survey that captures symptoms across five domains: sleep disturbance, physical suffering, emotional distress, daytime problems, and parent/caretaker concerns. With a Likert 7-point scale, caregivers rate the perceived frequency of 18 OSA-related problems ranging from 1 (none of the time) to 7 (all the time). Scores on each item are summed to produce a total score ranging from 18 to 126. Higher scores correspond to poorer sleep disordered breathing-related QOL, with a score greater than or equal to 60 signifying a clinically meaningful negative impact of sleep disordered breathing on QOL
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 193 | 186
change in score on a scale | -6.03 (14.59) | -15.77 (14.42)

9. Secondary Outcome: Change From Baseline to 12 Months in Body Mass Index (BMI) Percentile
Description: Body Mass Index (BMI) percentile, calculated from the average of triplicate in-clinic height/weight measurements. Percentiles calculated from Centers for Disease Control and Prevention (CDC) BMI-for-age charts.
Time Frame: 12 months
Population: All participants with 3 valid height and weight measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in percentile
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 188 | 187
change in percentile | 3.23 (13.31) | 5.09 (14.32)

10. Secondary Outcome: Change From Baseline to 12 Months in Mean Systolic and Diastolic Blood Pressures (mmHg) Percentile Scores.
Description: Mean of blood pressures measured in triplicate (to 1.0 mmHg) via automated oscillometric blood pressure cuff. Percentiles calculated respective to height, age and sex (PMID: 18230679).
Time Frame: 12 months
Population: All participants with 3 valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: Change in percentile
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 177 | 173
Change in percentile
  Systolic | 4.75 (31.4) | -4.5 (28.9)
  Diastolic: number analyzed (Participants) | 177 | 172
  Diastolic | 2.20 (20.79) | -4.87 (22.52)

11. Secondary Outcome: Change From Baseline to 12 Months in Average Heart Rate
Description: Average heart rate (beats per minute) calculated from overnight polysomnography
Time Frame: 12 months
Population: All participants with valid measurements at both baseline and 12-months are included
Measure: Mean (Standard Deviation); unit: change in avg bpm
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
Number analyzed (Participants) | 152 | 154
change in avg bpm | -1.80 (7.92) | -1.97 (7.68)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of the first consent through study completion, an average of 12 months with a maximum time frame of 425 days from consent.
Arm/Group | Watchful Waiting With Supportive Care | Early Adenotonsillectomy
All-Cause Mortality (participants affected / at risk) | 0/228 | 0/231
Serious Adverse Events (participants affected / at risk) | 9/228 | 13/231
Other Adverse Events (participants affected / at risk) | 112/228 | 103/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Watchful Waiting With Supportive Care (N=228) | Early Adenotonsillectomy (N=231)
Arm fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Broken ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Buckle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Closed fracture of clavicle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Closed fracture of unspecified part of fibula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Closed fracture of unspecified part of tibia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Croup (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Fracture of humerus, supracondylar closed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ketotic hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Physical abuse (Social circumstances) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postprocedural bleeding (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Watchful Waiting With Supportive Care (N=228) | Early Adenotonsillectomy (N=231)
Vomiting (Gastrointestinal disorders) | 15 (15) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 17 (18)
Streptococcal sore throat (Respiratory, thoracic and mediastinal disorders) | 30 (40) | 13 (14)
Stomach virus (Gastrointestinal disorders) | 16 (19) | 18 (19)
Postoperative pain (Injury, poisoning and procedural complications) | 0 (0) | 12 (14)
Influenza (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 19 (20)
Fever (General disorders) | 26 (34) | 16 (20)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 14 (16)
Ear infection (Ear and labyrinth disorders) | 25 (29) | 16 (21)
Common cold (Respiratory, thoracic and mediastinal disorders) | 27 (35) | 26 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT02562040/Prot_SAP_000.pdf